CLINICAL TRIAL: NCT04797299
Title: Prospective Evaluation of Breast-Conserving Surgery Alone in Low-Risk Ductal Carcinoma in Situ Defined by a Molecular Expression Assay Combined With Clinico-Pathological Features
Brief Title: Prospective Evaluation of Breast-Conserving Surgery Alone in Low-Risk Ductal Carcinoma in Situ (DCIS)
Acronym: ELISA
Status: Recruiting | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Other Study IDs: OCOG-2021-ELISA
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: DCIS
Keywords: Ductal Carcinoma in Situ; Breast Conserving Surgery; Oncotype DX DS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be used to determine Oncotype DX DCIS Score and subsequent testing for future correlative studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Arm Cohort: Evaluating the risk of Local Recurrence (LR) in a group of women postulated to be at low risk of LR following Breast Conserving Surgery alone defined by a combination of clinicopathological factors and Oncotype DX DCIS score.

SUMMARY:
To evaluate whether the combination of clinicopathological factors and the use of the Oncotype DX DCIS score can avoid radiation in women with low risk DCIS who have had breast conserving surgery (BCS)

DETAILED DESCRIPTION:
A prospective cohort study, conducted in Canada, to prospectively evaluate whether the combination of clinicopathological criteria and the Oncotype DX DCIS score can identify a group of women at very low risk of local recurrence following breast conserving surgery who do not require breast radiation therapy. We plan to screen 809 consenting women who will have their tumour tissue specimen sent to Exact Sciences to assess their DCIS score. We anticipate that 526 women will have an Oncotype DX DCIS score with a predicted 10-year risk of local recurrence ≤10%, these women will be enrolled and followed as part of the study.

At each centre, all patients with DCIS referred to radiation oncology will be documented. When a physician identifies an eligible patient, the patient will be approached by the referring physician or delegate to voluntarily provide informed consent to participate in this study. Consenting patients will be registered through the Ontario Clinical Oncology Group's (OCOG) web-based registration system. A two-step registration/enrollment process will be implemented.

Data related to the patient demographics, surgery details, tumour characteristics and ECOG performance will be collected. The patient's tumour specimen will be sent for analysis to Exact Sciences. The DCIS score results will be sent to the referring physician. OCOG will also receive the DCIS score results. Patients will be followed yearly up to 10 years. Bilateral mammograms and breast exams will be performed annually. The study data will be verified by source documentation.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient > 45 years of age with DCIS without microinvasion.
2. Tumour size ≤ 2.5cm.
3. Treated by BCS with clear resection margins ≥ 2 mm or no residual disease on re-excision.*

   * Patients with anterior margins and posterior margins ≥1 mm are eligible. Or if the dissection was confirmed to be taken to skin and down to fascia with no DCIS present at inked margins.
4. Oncotype DX DCIS score with a predicted 10-year risk of LR ≤10%.

Exclusion Criteria:

1. Multifocal DCIS.
2. History of any invasive breast cancer or non-invasive breast cancer in the ipsilateral breast.
3. Synchronous or previous invasive or non-invasive breast cancer.
4. Prior history of invasive cancer within the last 5 years, excluding non-melanoma skin cancers.
5. ECOG performance status ≥3.
6. Life expectancy <10 years.
7. Geographic inaccessibility for follow-up.

Min Age: 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort study conducted in Canada in women with a low risk DCIS following breast conserving surgery who are candidates for radiation.
  Eligibility status should be confirmed by the referring physician or delegate prior to enrollment. It is important that no exceptions are made to the eligibility criteria. Questions related to eligibility requirements and/or specific criteria should be addressed with OCOG prior to enrollment
Sampling Method: Probability Sample
Enrollment: 526 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2035-11-30 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral local recurrence (LR) | 5 Year
  Defined as recurrent invasive or in situ cancer in the ipsilateral breast

SECONDARY OUTCOMES:
Ipsilateral invasive local recurrence | 5 Year
  defined as time from study registration to time of recurrent invasive cancer in the ipsilateral breast
Breast cancer recurrence-free interval (RFI) | 5 Year
  defined as time from study registration to time of documented recurrent disease (ipsilateral breast (DCIS or invasive), regional, distant or death from breast cancer
Distant disease-free survival (DDFS) | 5 Year
  defined as time from study registration to distant recurrence
Disease-free survival (DFS) | 5 Year
  defined as time from registration to time of LR (DCIS or invasive), regional and distant recurrence, contralateral breast cancer, new primary (non-breast) and death from any cause
Overall survival (OS) | 5 Year
  defined as time from registration to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Rakovitch, M.D., Principal Investigator — Sunnybrook Research Institute, Sunnybrook Health Science; Tim Whelan, M.D, Principal Investigator — Juravinski Cancer Centre
Locations (24):
- Canada (24):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Abbotsford Centre, Abbotsford, British Columbia
  - BC Cancer - Centre for the North (Prince George), Prince George, British Columbia
  - BC Cancer - Fraser Valley Centre, Surrey, British Columbia
  - BC Cancer - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - QE II HSC - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Regional Cancer Care, Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Health Science Centre -Odette Cancer Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hôpital Charles Le Moyne (CISSS de la Montérégie-Centre), Greenfield Park, Quebec
  - CHUM - Centre Hospitalier de L'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec - Université Laval, Québec, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Mauricie- Centre-du-Québec (CIUSSS MCQ) - Trois-Rivières, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- See also: OCOG website accessed by clinical centres — http://www.ocog.ca